CLINICAL TRIAL: NCT03303768
Title: Antenatal Diagnosis of Coarctations of the Aorta. Prospective Observational Study.
Brief Title: Antenatal Diagnosis of Coarctations of the Aorta.
Acronym: CoA
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0477
Record Dates: First submitted 2017-09-28; First posted 2017-10-06 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Coarctation of Aorta
MeSH Terms: conditions — Aortic Coarctation | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women: Pregnant woman with suspected coarctation of isolated aorta or woman followed in the last 12 for suspected coarctation of the aorta isolated during pregnancy
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — Investigation of relevant ultrasound signs to improve the antenatal diagnosis of coarctation of the aorta by calculating the sensitivity and specificity of these different signs

SUMMARY:
Prenatal diagnosis of coarctation is difficult because the ductus arteriosus masks the isthmus narrowing. The problem lies in the fact that it is difficult to assert in utero diagnosis and to predict severity of neonatal symptomatology. However, it is essential to try to establish the diagnosis since it has been shown that the prenatal diagnosis improves survival and reduces morbidity.

ELIGIBILITY:
Inclusion Criteria:

* pregnant or having given birth in the last 12 months in one of the participating centers
* have had an ultrasound screening in the 2nd or 3rd trimester
* addressed or being addressed to the Pluridisciplinary Center for Prenatal Diagnosis for suspected coarctation of isolated aorta in front of: ventricular asymmetry at the aegis of the left ventricle or the large vessels at the aorta, discovered during a screening ultrasound second or third quarter.
* be able to understand and follow the ins and outs of the study
* Have been informed of the study and have not objected to it

Exclusion Criteria:

* Associated complex cardiac disease (transposition of large vessels, atrioventricular duct, right ventricle with double outlet) with the exception of inter ventricular communications
* Left ventricular hypoplasia
* Suspicion of interruption of the aortic arch

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Pregnant woman with suspected coarctation of isolated aorta or woman followed in the last 12 for suspected coarctation of the aorta isolated during pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-08-29 (Actual); Study Completion 2018-08-29 (Actual)

PRIMARY OUTCOMES:
Search for ultrasound risk factors associated with diagnosis coarctation of the aorta | 24h after birth
  Calculation of sensitivity, specificity and ROC (Receiver Operating Characteristic) curves of the different ultrasound parameters according to post-natal confirma-diagnosis of coarctation of the aorta in order to create a score to improve the antenatal diagnosis of coarctation the aorta.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Gynécologie Obstétrique Diagnostic Anténatal ; Hôpital Femme Mère enfant, Bron, France

IPD SHARING:
Plan to Share IPD: No